CLINICAL TRIAL: NCT05687669
Title: Comparison Between the Use of Phentolamine Versus Glyceryl Trinitrate for Their Effect on Renal Function in Pre-eclampsia Patients in ICU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ayman Abd El-Khalek Mohammed Glala, Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: obstetric Renal prophylaxis
Record Dates: First submitted 2022-12-07; First posted 2023-01-18 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Pre-Eclampsia; Complicating Pregnancy; Pre-eclampsia Aggravated
MeSH Terms: conditions — Pre-Eclampsia; Pregnancy Complications

STUDY DESIGN:
Intervention Model Description: Prospective study will be done in Assiut university hospital obstetric ICU, 2 groups will be examined and randomly assigned: group A using glyceryl trinitrate (GTN) to emergency control of blood pressure and group B using phentolamine infusion to control blood pressure. Each group consists of 85patients:
Who Masked: Participant
Masking Description: Group(A): Glyceryl trinitrate (GTN) is labelled with "Drug A" on syringe pump. Group(B): Phentolamine is labelled with "Drug B" on syringe pump.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group GTN (Experimental): Glyceryl trinitrates (GTN) is infused to patients with severe hypertensive preeclampsia till oral anti-hypertensives and Magnesium sulfate loadings lower blood pressure
  Interventions: Drug: Glyceryl trinitrate vs phentolamine for prophylaxis against renal impairment
- Group Phentolamine (Experimental): Phentolamine is infused to patients with severe hypertensive preeclampsia till oral anti-hypertensives and Magnesium sulfate loadings lower blood pressure
  Interventions: Drug: Glyceryl trinitrate vs phentolamine for prophylaxis against renal impairment

INTERVENTIONS:
Drug: Glyceryl trinitrate vs phentolamine for prophylaxis against renal impairment — Glyceryl trinitrate vs phentolamine for prophylaxis against renal impairment

SUMMARY:
Severe pre-eclamptic toxemia has a high incidence of renal complications. Rapid diagnosis and termination of pregnancy are still the gold standard main treatment for pre-eclampsia. Rapid control of blood pressure showed to provide protection against many adverse effects of preeclampsia as intracranial hemorrhage, subcapsular hepatic hematoma and acute kidney injury (AKI).

In Assiut university hospital ICU regimen, glyceryl trinitrate (GTN) was used primarily for this purpose. But it was accused in many cases as a cause for AKI without any other organ damage along with the severe preeclampsia disease. Some previous studies supported this assumption as , Ying-Hsuan .T. et.,al during their study of GTN on renal outcome during cardiopulmonary bypass in cardiac surgery. Phentolamine infusion is a new rising alternative for an old drug with a high safety profile.

In this research protocol the researchers will study comparative effect of glyceryl trinitrate (GTN) versus phentolamine on renal outcome in severe pre-eclampsia patients during their stay in obstetric ICU.

ELIGIBILITY:
Inclusion Criteria:

* Severe preeclampsia defined by presentation of 2 or more of the following criteria:

  1. Blood pressure more than 160/100
  2. Proteinuria
  3. Pitting edema
  4. With or without organ dysfunctions

Exclusion Criteria:

1. Patient relatives' refusal
2. Recent active internal hemorrhage
3. Chronic renal impairment or failure on dialysis for any other etiology

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — only in preeclampsia patients which is complicating pregnancy in females
Enrollment: 170 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-06-12 (Actual)

PRIMARY OUTCOMES:
kidney function tests | 96 hours after intervention
  creatinine in micromoles per liter and urea in millimole per liter

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university faculty of medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided